CLINICAL TRIAL: NCT07036627
Title: Evaluation of the Intestinal Microbiota in Pediatric Patients Treated With Proton Pump Inhibitors: A Prospective Longitudinal Study
Brief Title: Intestinal Microbiota After PPI Treatment
Acronym: PPI
Status: Not yet recruiting | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Ruggiero Francavilla, Prof Ruggiero Francavilla, University of Bari
Other Study IDs: PPI
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Proton Pump Inhibitors; Human Gastrointestinal Tract; Gastroesophageal Reflux Disease
Keywords: PPI; GERD; microbiota; gastroesophageal reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PPI: PPI
  Interventions: Other: study of microbiota

INTERVENTIONS:
Other: study of microbiota — * Drug: Esomeprazole, a proton pump inhibitor commonly used in pediatric gastroenterology.
  * Administration: Oral, once daily, 30 minutes before meals.
  * Dosage: Personalized dosing according to body weight, with an average of approximately 0.6 mg/kg/day.
  * Treatment duration: Minimum 45 days, maximum 60 days.
  * Comparator: None. This is a within-subject design; each participant serves as their own control with baseline samples (t0) compared to follow-up (t1-t2).
  * Monitoring: Adherence to therapy and sample collection timeline will be verified during scheduled clinical follow-up.

SUMMARY:
This clinical study aims to investigate the effects of short-term treatment with proton pump inhibitors (PPIs) on the gut microbiota of pediatric patients. PPIs are among the most frequently prescribed medications in children and adolescents for the management of acid-related disorders, such as gastroesophageal reflux disease (GERD). However, emerging evidence suggests that these medications may have unintended consequences on the delicate ecosystem of beneficial microorganisms residing in the human gastrointestinal tract.

The intestinal microbiota plays a pivotal role in modulating immune responses, supporting nutrient metabolism, and maintaining the integrity of the gut barrier. Disruption of this microbial balance-known as dysbiosis-has been associated with several health conditions, including infections, allergies, obesity, and chronic inflammation. In adults, long-term PPI use has been linked to microbiota alterations, but data in the pediatric population remain limited and inconclusive.

To address this gap, our prospective longitudinal study will recruit pediatric patients prescribed PPI therapy for clinical indications. Stool samples will be collected at four time points: prior to PPI administration, during treatment, and at two follow-up stages post-cessation. Using 16S rRNA gene sequencing, we will profile changes in microbial diversity and abundance over time.

The results will offer insight into whether short-term PPI exposure in children leads to significant, lasting changes in gut microbiota composition or diversity. Such information may ultimately inform prescribing practices, support personalized therapeutic strategies, and help mitigate potential risks associated with microbiota disruption during childhood-a critical period for microbial and immune system development.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children and adolescents aged between 6 months and 17 years at the time of enrollment.
* Clinical indication for proton pump inhibitor therapy, including but not limited to gastroesophageal reflux disease, esophagitis, or functional dyspepsia.
* Willingness and ability of the child and their caregivers to comply with all study procedures, including collection of fecal samples at scheduled time points.
* Written informed consent obtained from a parent or legal guardian; assent obtained from the child, when age-appropriate, in accordance with local regulations and ethical standards.

Exclusion Criteria:

* Use of systemic antibiotics, antifungals, or probiotics within 30 days prior to the start of the study or during the observation period.
* Incomplete or improperly handled stool sample collection, or failure to adhere to protocol-defined sampling windows.
* Known diagnosis of primary immunodeficiency, inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis), or celiac disease.
* Any condition that, in the opinion of the investigator, may interfere with the integrity of the study or pose additional risks to the participant.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Population with GERD
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-06 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in microbiota | 60 days from baseline
  * Definition: Change in the relative abundance of key bacterial families (Streptococcaceae, Ruminococcaceae, Clostridiales, etc.) from t0 to t1.
  * Methodology: High-throughput 16S rRNA gene sequencing (regions V3-V4) using the Illumina MiSeq platform; taxonomic assignment via the SILVA reference database.
  * Justification: These bacterial families have been previously associated with dysbiosis and PPI-related shifts in microbial composition.

SECONDARY OUTCOMES:
Microbial diversity | 60 days from baseline.
  * Alpha-diversity: Within-sample microbial diversity measured by Shannon's entropy and Chao1 richness estimator.
  * Beta-diversity: Between-sample differences using Bray-Curtis dissimilarity; visualized via principal coordinates analysis (PCoA).
  * Differential abundance: Identification of statistically enriched or depleted taxa using LEfSe (Linear Discriminant Analysis Effect Size).
  * Clinical correlation: Incidence of gastrointestinal (e.g., diarrhea, abdominal pain) and respiratory symptoms (e.g., cough, wheezing) reported during or after therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatria Trambusti, Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mitre E, Susi A, Kropp LE, Schwartz DJ, Gorman GH, Nylund CM. Association Between Use of Acid-Suppressive Medications and Antibiotics During Infancy and Allergic Diseases in Early Childhood. JAMA Pediatr. 2018 Jun 4;172(6):e180315. doi: 10.1001/jamapediatrics.2018.0315. Epub 2018 Jun 4. PMID 29610864
- [Background] Simakachorn L, Tanpowpong P, Chanprasertyothin S, Thongpradit S, Treepongkaruna S. Gut Microbiota Characteristics in Children After the Use of Proton Pump Inhibitors. Turk J Gastroenterol. 2021 Jan;32(1):70-75. doi: 10.5152/tjg.2020.20245. PMID 33893768
- [Background] Raisanen L, Viljakainen H, Kolho KL. Exposure to proton pump inhibitors is associated with the development of pediatric autoimmune diseases. Front Pediatr. 2023 Mar 27;11:1157547. doi: 10.3389/fped.2023.1157547. eCollection 2023. PMID 37051434
- [Background] Levy EI, Hoang DM, Vandenplas Y. The effects of proton pump inhibitors on the microbiome in young children. Acta Paediatr. 2020 Aug;109(8):1531-1538. doi: 10.1111/apa.15213. Epub 2020 Mar 18. PMID 32027402
- [Background] Zhang YJ, Connearney S, Hester L, Du M, Catacora A, Akkara A, Wen A, Bry L, Alm EJ, Rosen R. Longitudinal Microbiome Changes in Children Exposed to Proton Pump Inhibitors. Clin Transl Gastroenterol. 2024 Sep 1;15(9):e1. doi: 10.14309/ctg.0000000000000703. PMID 38624107
- [Background] Liu C, Bach TR, Farrell PM, Pavelec D, Antos NJ, Rock MJ, Asfour F, Howenstine M, Gaffin JM, Lai HJ. Impact of acid blocker therapy on growth, gut microbiome, and lung disease in young children with cystic fibrosis. J Pediatr Gastroenterol Nutr. 2024 Dec;79(6):1124-1133. doi: 10.1002/jpn3.12389. Epub 2024 Oct 28. PMID 39465618